CLINICAL TRIAL: NCT06980298
Title: Toxoplasma Gondii Seroprevalence Among Children With Some Neuropsychiatric Disorders in Sohag Governorate, Egypt
Brief Title: Toxoplasma Gondii Seroprevalence Among Children With Some Neuropsychiatric Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Abdelhameed Elsayed, Alaa Abd Elhamid Elsayed Mohamed, Sohag University
Other Study IDs: Soh-Med--25-4-04MS
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Toxoplasmosis in Neuropsychiatric Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: 45 blood samples will be collected from children have either epilepsy or ADHD. Approximately 3 ml venous blood will be collected from each child by venipuncture, under sterile conditions.
- Control group: 45 blood samples will be collected from matched children for age and gender, served as control.
  Approximately 3 ml venous blood will be collected from each child by venipuncture, under sterile conditions.

SUMMARY:
Toxoplasma gondii is recognized as being involved in the etiology of various psychotic disorders including epilepsy and ADHD (Markovitz et al.,2015).

There are many explanations for such associations between toxoplasmosis and neurological disorders which include many anatomical and neurotransmitter-related changes. Toxoplasmosis may cause alterations in neurotransmitter levels like serotonin, noradrenaline, glutamate, nitric oxide and gamma aminobutyric acid, increase in the levels of proinflammatory cytokines and modulate the dopaminergic signaling (Babaie et al., 2017). The behavioral changes produced by the cyst formation in the brain tissue may also related to the localization of the cyst within specific parts of the brain and this is assumed to be one of the main causes of epilepsy in toxoplasmosis. Moreover, tachyzoites may invade the brain tissues and excite brain cells especially neurons, microglia and astrocytes. Additionally, the presence of Toxoplasma in brain evokes inflammatory response and stimulate immune system to produce antibodies with increase in proinflammatory cytokines. Interestingly, some studies described that many host genes and proteins could be affected by Toxoplasma, signifying its involvement in many genetic disorders including neuropsychiatric diseases.The current study aimed to assess the seroprevalence of anti-Toxoplasma IgM and IgG antibodies among children with some neuropsychiatric disorders (Epilepsy and ADHD) in Sohag governorate, Egypt.

ELIGIBILITY:
Inclusion criteria: Children with neuropsychiatric disorders (epilepsy,ADHD). Exclusion criteria: Children with history of neurosurgery, head injury or trauma, neoplastic or autoimmune diseases, or receiving immunosuppressant or systemic corticosteroid, and those with possible neurological infection.

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 90 children will be collected from children ,45 of them have either epilepsy or ADHD and another matched 45 children for age and gender, served as control.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Comparison between incidence of Toxoplasma gondii in children with neuropsychiatric disorders and children without neuropsychiatric disorders | 6 months

SECONDARY OUTCOMES:
Prevalence of Toxoplasma gondii in children with neuropsychiatric disorders | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided